CLINICAL TRIAL: NCT02801214
Title: Effects of Recreational Cannabis Use on Brain Activation Patterns Associated With Emotional Processes
Brief Title: Emotional Brain Processes in Recreational Cannabis Users
Status: Completed | Type: Observational
Sponsor: University of Electronic Science and Technology of China (Other)
Collaborators: German Research Foundation (Other); University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Prof. Dr. rer. nat. Benjamin Becker, University of Electronic Science and Technology of China
Other Study IDs: ART_Can_02
Record Dates: First submitted 2016-06-11; First posted 2016-06-15 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Recreational Cannabis Use
Keywords: cannabis; fMRI; emotion
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Recreational Cannabis Use: ages 18-40
  Interventions: Other: fMRI
- Healthy control subjects: socio-demographically matched
  Interventions: Other: fMRI

INTERVENTIONS:
Other: fMRI

SUMMARY:
This fMRI study investigates neural correlates of emotion regulation, emotion processing and craving in recreational cannabis users.

ELIGIBILITY:
Inclusion Criteria:

* Recreational cannabis use
* 72 hours of abstinence

Exclusion Criteria:

* neurological disorders
* psychiatric disorders according to DSM-4

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Recreational male cannabis users
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
fMRI neural correlates of emotional brain processes in recreational cannabis users after 72 hours of abstinence | one time point = fMRI assessment after 72 hours of abstinence
  Activation patterns in brain regions known to be involved in emotional processing and to be altered by cannabis use (e.g. striatum, prefrontal cortex, insula, ACC)

SECONDARY OUTCOMES:
Ratings of subjective experience (affect, craving) | one time point = during fMRI assessment after 72 hours of abstinence